CLINICAL TRIAL: NCT00653042
Title: A Pilot, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Nesiritide Infusion, Initiated Post-Induction of Anesthesia, in the Management of Coronary Artery Bypass Graft (CABG) Patients Requiring CardioPulmonary Bypass (CPB)
Brief Title: Clinical Study to Evaluate Nesiritide in Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery A014 / NAPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR003352; NCT00090792 (obsolete NCT alias)
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Coronary Artery Bypass Surgery; Coronary Heart Disease; Coronary Artery Bypass Grafting; Cardiopulmonary Bypass; Ischemic Heart Disease; Congestive Heart Failure
Keywords: Myocardial Ischemia; kidney failure; CABG; cardiopulmonary bypass (CPB) pump; Coronary Artery Bypass Surgery; heart surgery; nesiritide; Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia; Heart Failure; Renal Insufficiency | interventions — Natriuretic Peptide, Brain

INTERVENTIONS:
Drug: Nesiritide

SUMMARY:
The purpose of this study is to assess the effects of nesiritide compared to placebo when given with standard of care therapies, on kidney function, heart function and the need of other treatments in heart failure patients undergoing heart bypass graft surgery that requires the use of a cardiopulmonary bypass machine (CPB pump or heart-lung machine).

DETAILED DESCRIPTION:
In coronary heart disease (CHD), the coronary arteries become clogged with calcium and fatty deposits. The deposits, called plaques, narrow the arteries that carry blood to the heart muscle and could cause ischemic heart disease (too little blood and oxygen reaching the heart muscle). Coronary Artery Bypass Graft (CABG) surgery is a treatment option for ischemic heart disease. CABG surgery is surgery to create new routes for blood to flow around narrowed and blocked arteries so that the heart muscle will receive needed oxygen and nutrients. Acute kidney injury is a serious risk of CABG surgery while on CPB pump (heart-lung machine), which could result from ischemia during and following surgery. This study is a double-blind (neither the patient nor the doctor knows whether the patient is assigned to receive study drug or placebo), randomized (assigned to treatment by chance), placebo-controlled (study drug results compared to placebo results) study to determine the effectiveness of nesiritide compared to placebo when given to HF patients undergoing CABG surgery requiring the use of a CPB pump . Patients will be enrolled into the study until 250 patients have received study drug or placebo. Patients will be randomized to one of two treatment groups in a 1:1 ratio (nesiritide plus standard care: placebo plus standard care) within each site. Study medication administration will be initiated after measurement of qualifying baseline hemodynamics and prior to chest incision. Nesiritide or placebo will be administered as a continuous IV infusion at a rate of 0.01 mcg/kg/min for a minimum of 24 hours and a maximum of 96 hours. Patients will be followed through 30 days from start of study drug. All patients may receive additional standard care medications including inotropes, pressors, vasopressin, antiarrhythmics, diuretics, nitrates, and nitric oxide as needed. Patient safety will be monitored throughout the study through physical exams, vital signs (heart rate, blood pressure, respiratory rate, and temperature), blood tests, and side effects. A follow-up communication 180 days after the start of study drug was implemented to collect mortality data. The patients assigned to the nesiritide group will receive a continuous I.V. infusion at 0.010 mcg/kg/min of nesiritide for at least 24 hours and could be extended to up to 96 hours. The patients assigned to the placebo group will receive matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* NYHA class II-IV CHF
* Presenting for CABG with or without mitral valve repair or replacement procedure
* Planned utilization of CPB
* Documentation of left ventricular ejection fraction (LVEF) less than or equal to 40% measured by nuclear scan, echocardiogram (ECHO), or ventriculogram, within 90 days prior to surgery.

Exclusion Criteria:

* Planned aortic valve replacement or repair
* Ongoing or chronic dialysis (either hemodialysis or continuous ambulatory peritoneal dialysis)
* Restrictive or obstructive cardiomyopathy, constrictive pericarditis, pericardial tamponade, or other conditions in which cardiac output is dependent on venous return
* Documented or suspected low cardiac filling pressures
* Any known congenital heart disease
* Known allergic reaction or sensitivity to nesiritide or excipients
* Females of childbearing potential with a positive serum pregnancy test, and nursing mothers
* Treated with investigational drug or device within last 30 days
* documented fever (>101 degrees F) within 72 hours of surgery
* WBC > 15,000/mm3 within 72 hours of surgery
* Documented bacterial/fungal/viral infection requiring administration of IV antibiotics within 7 days before surgery
* Pulmonary disease (COPD, asthma or other condition) that required inpatient medical or surgical treatment within 60 days before surgery. Treatment exclusion criteria (obtained after anesthesia induction and before chest incision prior to the start of study drug) include: mean pulmonary artery pressure consistently < or equal to 15mmHg
* central venous pressure consistently < 6 mmHg
* and systolic blood pressure consistently < 90 mmHg. Use of open-label nesiritide within 48 hours of study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2004-03; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline serum creatinine, total inotrope/vasopressor/vasodialator use during first 24 hours, average change from baseline of mean PAP for 24 hours from study start or after removal of catheter and 24-hour urine output after ICU/CCU admission

SECONDARY OUTCOMES:
Time to extubation, Time to discharge from ICU/CCU and hospital, Time on CPB, Adverse Events, and Change from baseline in hemodynamic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- See also: Clinical study to evaluate nesiritide in patients undergoing Coronary Artery Bypass Graft (CABG) surgery A014 / NAPA — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=954&filename=CR003352_CSR.pdf